CLINICAL TRIAL: NCT00000566
Title: Prospective Investigation of Pulmonary Embolism Diagnosis (PIOPED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Diagnostic
Other Study IDs: 204
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2002-06

CONDITIONS: Lung Diseases; Pulmonary Embolism
MeSH Terms: conditions — Lung Diseases; Pulmonary Embolism | interventions — Ventilation-Perfusion Ratio; Cerebral Angiography

INTERVENTIONS:
Procedure: ventilation-perfusion ratio
Procedure: angiography

SUMMARY:
To evaluate the sensitivity and specificity of two major, widely used technologies, radionuclear imaging (ventilation-perfusion scanning) and pulmonary angiography, for the diagnosis of pulmonary embolism.

DETAILED DESCRIPTION:
BACKGROUND:

In 1983, reliable data on the incidence of pulmonary embolism in the adult population and in groups identified at risk were not available because the sensitivity and specificity of the diagnostic procedures had not been determined. Estimates suggested there were about half a million episodes of pulmonary embolism in hospitalized patients each year in the United States. Deaths attributable to pulmonary embolism would be expected in about one third of these patients if left untreated.

The clinical diagnosis of pulmonary embolism was subject to a high frequency of false positives and false negatives. The most definitive diagnostic procedure was pulmonary angiography, an invasive, expensive procedure which was not without risk. It required specialized equipment and highly trained personnel both for performance and for interpretation. Therefore, it was used to diagnose pulmonary embolism only in the major medical centers. Another technique utilized as a method to diagnose pulmonary embolism involved a combination of perfusion and ventilation scanning; this method was only minimally invasive. A normal perfusion scan was thought to be of considerable value because it essentially excluded the diagnosis of pulmonary embolism. In selected patient populations, abnormal perfusion scans combined with normal ventilation scans were of substantial help in diagnosis.

Although there had been no acceptable validation of the use of perfusion scans in the diagnosis of pulmonary embolism, thousands of patients had been evaluated for pulmonary embolism based on perfusion scanning often using methods of imaging now considered to be inadequate. In the early 1980s, clinical practice interpreted a negative perfusion scan as overwhelming evidence against the presence of pulmonary emboli. This interpretation had not been adequately tested either in a prospective study or by long-term follow-up of patients to determine clinical outcome. With regards to positive perfusion scans, there were data to suggest that as many as two-thirds of positive perfusion scans could not subsequently be confirmed by pulmonary angiography. Prospective studies in which timely angiograms using selective injections and improved imaging techniques were needed to evaluate the usefulness of positive perfusion scans.

Phase I was initiated in September 1983. Protocols developed during Phase I underwent independent assessment review in April 1984 and were reviewed and approved by the May 1984 National Heart, Lung, and Blood Advisory Council. Recruitment and intervention started in January 1985 and ended in September 1986. Follow-up was completed on September 30, 1987.

DESIGN NARRATIVE:

Patients suspected of pulmonary embolism underwent a ventilation-perfusion scan. Patients with an abnormal perfusion scan underwent angiography. All patients were followed for one year.

ELIGIBILITY:
Men and women suspected of having a pulmonary embolism and who met the criteria to undergo angiography.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1983-09; Study Completion 1989-12

CONTACTS AND LOCATIONS:
Overall Officials: Abass Alavi — University of Pennsylvania; Richard Greenspan — Yale University; Charles Hales — Massachusetts General Hospital; Herbert Saltzman — Duke University; Paul Stein — Henry Ford Hospital; John Weg — University of Michigan

REFERENCES:
- [Background] Henry JW, Stein PD, Gottschalk A, Raskob GE. Pulmonary embolism among patients with a nearly normal ventilation/perfusion lung scan. Chest. 1996 Aug;110(2):395-8. doi: 10.1378/chest.110.2.395. PMID 8697840
- [Background] Gottschalk A, Stein PD, Henry JW, Relyea B. Can pulmonary angiography be limited to the most suspicious side if the contralateral side appears normal on the ventilation/perfusion lung scan? Data from PIOPED. Prospective Investigation of Pulmonary Embolism Diagnosis. Chest. 1996 Aug;110(2):392-4. doi: 10.1378/chest.110.2.392. PMID 8697839
- [Background] Tissue plasminogen activator for the treatment of acute pulmonary embolism. A collaborative study by the PIOPED Investigators. Chest. 1990 Mar;97(3):528-33. doi: 10.1378/chest.97.3.528. PMID 2106408
- [Background] PIOPED Investigators. Value of the ventilation/perfusion scan in acute pulmonary embolism. Results of the prospective investigation of pulmonary embolism diagnosis (PIOPED). JAMA. 1990 May 23-30;263(20):2753-9. doi: 10.1001/jama.1990.03440200057023. PMID 2332918
- [Background] Bone RC. Ventilation/perfusion scan in pulmonary embolism. 'The Emperor is incompletely attired'. JAMA. 1990 May 23-30;263(20):2794-5. No abstract available. PMID 2185372
- [Background] Stein PD, Gottschalk A, Saltzman HA, Terrin ML. Diagnosis of acute pulmonary embolism in the elderly. J Am Coll Cardiol. 1991 Nov 15;18(6):1452-7. doi: 10.1016/0735-1097(91)90674-x. PMID 1939945
- [Background] Stein PD, Alavi A, Gottschalk A, Hales CA, Saltzman HA, Vreim CE, Weg JG. Usefulness of noninvasive diagnostic tools for diagnosis of acute pulmonary embolism in patients with a normal chest radiograph. Am J Cardiol. 1991 May 15;67(13):1117-20. doi: 10.1016/0002-9149(91)90875-l. PMID 2024602
- [Background] Stein PD, Coleman RE, Gottschalk A, Saltzman HA, Terrin ML, Weg JG. Diagnostic utility of ventilation/perfusion lung scans in acute pulmonary embolism is not diminished by pre-existing cardiac or pulmonary disease. Chest. 1991 Sep;100(3):604-6. doi: 10.1378/chest.100.3.604. PMID 1889240
- [Background] Stein PD, Terrin ML, Hales CA, Palevsky HI, Saltzman HA, Thompson BT, Weg JG. Clinical, laboratory, roentgenographic, and electrocardiographic findings in patients with acute pulmonary embolism and no pre-existing cardiac or pulmonary disease. Chest. 1991 Sep;100(3):598-603. doi: 10.1378/chest.100.3.598. PMID 1909617
- [Background] Stein PD, Saltzman HA, Weg JG. Clinical characteristics of patients with acute pulmonary embolism. Am J Cardiol. 1991 Dec 15;68(17):1723-4. doi: 10.1016/0002-9149(91)90339-m. No abstract available. PMID 1746481
- [Background] Stein PD, Athanasoulis C, Greenspan RH, Henry JW. Relation of plain chest radiographic findings to pulmonary arterial pressure and arterial blood oxygen levels in patients with acute pulmonary embolism. Am J Cardiol. 1992 Feb 1;69(4):394-6. doi: 10.1016/0002-9149(92)90240-y. PMID 1734655
- [Background] Quinn DA, Thompson BT, Terrin ML, Thrall JH, Athanasoulis CA, McKusick KA, Stein PD, Hales CA. A prospective investigation of pulmonary embolism in women and men. JAMA. 1992 Oct 7;268(13):1689-96. PMID 1527878
- [Background] Carson JL, Kelley MA, Duff A, Weg JG, Fulkerson WJ, Palevsky HI, Schwartz JS, Thompson BT, Popovich J Jr, Hobbins TE, et al. The clinical course of pulmonary embolism. N Engl J Med. 1992 May 7;326(19):1240-5. doi: 10.1056/NEJM199205073261902. PMID 1560799
- Available data/document: Individual Participant Data Set: PIOPED — http://biolincc.nhlbi.nih.gov/studies/pioped/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/pioped/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/pioped/